CLINICAL TRIAL: NCT04539522
Title: A Prospective Clinical Study on the Efficacy of a Three-dimensionally Corrective Exercise Therapy for Scoliosis
Brief Title: Efficacy of a Three-dimensionally Corrective Exercise Therapy for Scoliosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XHEC-SHHDC-2021-009-2
Record Dates: First submitted 2020-08-28; First posted 2020-09-07 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Idiopathic Scoliosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three-dimensionally corrective exercise for scoliosis (Experimental): Experimental group will perform three-dimensionally corrective exercise for scoliosis for a 60-min period for 1-2 times a week under the guidance of physical therapist in an outpatient clinic, and a 40-min period per day under the supervision of the parents at home.For moderate patients, additional brace treatment for more than 22 hours a day.The treatment regimens lasted for 12 months.
  Interventions: Behavioral: Three-dimensionally corrective exercise for scoliosis
- Conventional exercise (Active Comparator): Control subjects will perform conventional exercise for a 60-min period for 1-2 times a week under the guidance of physical therapist in an outpatient clinic, and a 40-min period per day under the supervision of the parents at home. For moderate patients, additional brace treatment for more than 22 hours a day.The treatment regimens lasted for 12 months.
  Interventions: Behavioral: Conventional exercise

INTERVENTIONS:
Behavioral: Three-dimensionally corrective exercise for scoliosis — Three-dimensionally corrective exercise for scoliosis is based the theory of physiotherapeutic scoliosis specific exercises, which focus on 3-dimension self-correction and consists of two parts:1)outpatient treatment including stretching, three-dimensional auto-correction(combine with specific breathing mode, isometric training to correct abnormal spinal physiological curvatures in sagittal plane, and accompany with wedge pad to modify humpback, waist asymmetry, pelvic rotation in horizontal. While in coronal plane, longitudinal axial stretching, pelvic adjustments will be conducted to reduce the lateral curvature.), balance and stability training, combined with manual fascia relaxation therapy, and and breathing training; 2)family rehabilitation: combines self-correcting gymnastics with daily posture management, etc., forming the individual exercise approach for each patient.
  Arms: Three-dimensionally corrective exercise for scoliosis
Behavioral: Conventional exercise — Conventional exercise consists a series of spine exercises focusing on core strength training.
  Arms: Conventional exercise

SUMMARY:
Idiopathic scoliosis (AIS) is one of the most prevalent spinal deformity that may progress sharply during growth. It is recommended that the physiotherapeutic scoliosis-specific exercises should be the first step to treat idiopathic scoliosis to prevent/limit progression of the deformity. Three-dimensionally corrective exercise for scoliosis is based the theory of physiotherapeutic scoliosis specific exercises, which focuses on 3-dimension self-correction and consists of two parts:1)outpatient treatment including stretching, three-dimensional self-correction, balance and stability training, combined with manual fascia relaxation therapy, and and breathing training; 2)family rehabilitation: combines self-correcting gymnastics with daily posture management, etc., forming the individual exercise approach for each patient. Nevertheless, the evidence concerning three-dimensionally corrective exercise for scoliosis is inadequate. Therefore, the objective of this study is to determine the effect of three-dimensionally corrective exercise intervention on the change of Cobb angle, trunk rotation, sagittal profile, lung function, exercise endurance and health related quality-of-life, compared to conventional exercise therapy for patients with mild and moderate AIS.

Informed consent will be obtained from each patient and one of their parents prior to inclusion. Eligible subjects will be divided into two groups(experimental group or control group) according to their wishes. Subjects in experimental group will perform three-dimensionally corrective exercise for scoliosis (moderate patients combined with a brace) and those in the control group will receive conventional exercise therapy (moderate patients combined with a brace).

Blinded assessments at baseline and immediately post 12-month intervention will include radiographic measurement, trunk rotation, sagittal profile, lung function, exercise endurance and health related quality-of-life.

DETAILED DESCRIPTION:
Idiopathic scoliosis (AIS) is one of the most prevalent spinal deformity that may progress sharply during growth. According to the severity of the curve, the major treatment approaches for patient with AIS include exercises, bracing and surgery, to correct, prevent or stop the progression of the deformity.In North America, Scoliosis Research Society (SRS) has been published the standard of care for AIS: patients with curves between 10 and 25° should be observation who are still growing. While in the Europe, the International Scientific Society on Scoliosis Orthopaedic and Rehabilitation Treatment (SOSORT) has recommended that the physiotherapeutic scoliosis-specific exercises should be the first step to treat idiopathic scoliosis to prevent/limit progression of the deformity. Three-dimensionally corrective exercise for scoliosis is based the theory of physiotherapeutic scoliosis specific exercises, which focuses on 3-dimension self-correction and consists of two parts:1)outpatient treatment including stretching, three-dimensional self-correction, balance and stability training, combined with manual fascia relaxation therapy, and and breathing training; 2)family rehabilitation: combines self-correcting gymnastics with daily posture management, etc., forming the individual exercise approach for each patient. Nevertheless, the evidence concerning three-dimensionally corrective exercise for scoliosis is inadequate. Therefore, the objective of this study is to determine the effect of three-dimensionally corrective exercise intervention on the change of Cobb angle, trunk rotation, sagittal profile, lung function, exercise endurance and health related quality-of-life, compared to conventional exercise therapy for patients with mild and moderate AIS.

The present study is a single-center prospective non-randomised controlled trial conducted at the department of rehabilitation medicine, Xinhua Hospital affiliated to Shanghai Jiao Tong University School of Medicine. The demographic data (height, weight), menarche status for the girls, family history, will be recorded by the physician.

Informed consent will be obtained from each patient and one of their parents prior to inclusion. Eligible subjects will be assigned by a 1:1 allocation ratio either to the experimental group, in which they will perform three-dimensionally integrated exercise for scoliosis, or the control group, in which they will receive the standard of care with observation according to the Scoliosis Research Society criteria. Blinded assessments at baseline and immediately post 12-month intervention will include radiographic measurement, trunk rotation, sagittal profile, lung function, exercise endurance and health related quality-of-life.

ELIGIBILITY:
Inclusion Criteria(meet all the following conditions):

1. Age between 8-16;
2. Definitely diagnosed as IS;
3. Patients with Cobb angle greater than or equal to 10° and less than 45°.

Exclusion Criteria(at least meet one of the following conditions):

1. Scoliosis caused by congenital, postural, neuromuscular or other diseases (such as neurofibromatosis, Marfan syndrome, bone dysplasia, metabolic or endocrine diseases, etc.);
2. Patients suffering from mental illness or rheumatic disease;
3. Patients with insufficient understanding ability to understand and complete the treatment plan;
4. Patients with exercise contraindications who cannot tolerate exercise therapy;
5. Patients with poor treatment compliance or refusal to treat;
6. Patients with a history of rehabilitation or surgery before the first visit;
7. Patients with apical vertebrae at T7 and above, or patients with mature bones.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 172 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Change of Cobb angle | up to 12 months
  It is recommended that curve magnitude of scoliosis is measured using the Cobb method. The Cobb angle will be measured on the standing frontal radiograph according to the Cobb method by the physician specializing in the treatment of scoliosis.

SECONDARY OUTCOMES:
Angle of trunk rotation | up to 12 months
  The angle of trunk rotation will be measured with a Scoliometer. Patients will be asked to bend forward, and the physician will measure the angle of trunk rotation using the Scoliometer.
Sagittal index | up to 12 months
  The Sagittal index (SI) is the sum of plumbline distances from C7 and L3. When SI<60mm,it is considered to be flat black; 60-90mm is in the normal range; >90 mm is considered to kyphosis.
Forced vital capacity | up to 12 months
  Forced vital capacity (FVC) is an established measure of pulmonary function.
Forced expiratory volume in first second | up to 12 months
  Forced expiratory volume in first second is an established measure of pulmonary function.
Peak oxygen uptake | up to 12 months
  Peak oxygen uptake is recognised as the best expression of exercise endurance and will be measured by cardiopulmonary exercise testing.
Scoliosis Research Society-22 (SRS-22) questionnaire score | up to 12 months
  Scoliosis Research Society-22 (SRS-22) questionnaire was designed for patients with scoliosis specially , which consists of 22 items with 5 dimensions: function/activity, pain, self-Image, mental health, and satisfaction with treatment. The higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Du, Ph.D, Principal Investigator — Xin Hua Hospital,Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xin Hua Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhou X, Li X, Wu Q, Liang J, Guo H, Jin M, Zhu X, Du Q. Three-dimensional corrective exercise therapy for idiopathic scoliosis: study protocol for a prospective non-randomized trial. BMC Musculoskelet Disord. 2022 Feb 5;23(1):118. doi: 10.1186/s12891-022-05057-7. PMID 35123460